CLINICAL TRIAL: NCT03409081
Title: Early Access Program (EAP) of Gilteritinib (ASP2215) in Patients With FMS-like Tyrosine Kinase 3 (FLT3) Mutated Relapsed or Refractory Acute Myeloid Leukemia (AML) or With FLT3-Mutated AML in Complete Remission (CR) With Minimal Residual Disease (MRD)
Status: No longer available | Type: Expanded Access
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2215-CL-9200
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Acute Myeloid Leukemia (AML); FMS-like Tyrosine Kinase-3 (FLT3) Mutations
Keywords: Expanded Access; FMS-like Tyrosine Kinase 3; Acute Myeloid Leukemia (AML); gilteritinib; ASP2215
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: gilteritinib — oral
  Other Names: ASP2215

SUMMARY:
The purpose of this study is to provide expanded access to gilteritinib (ASP2215) for patients with FMS-like tyrosine kinase 3 (FLT3)-mutated relapsed or refractory acute myeloid leukemia (AML) or with FLT3-mutated AML in composite complete remission (CRc: [complete remission (CR), complete remission with incomplete hematologic recovery (CRi), complete remission with incomplete platelet recovery (CRp)]) with minimal residual disease (MRD) without access to comparable or alternative therapy.

DETAILED DESCRIPTION:
This treatment protocol is being conducted while phase 3 gilteritinib (ASP2215) studies are ongoing in FLT3-mutated AML patients.

Patients will be administered treatment over 28-day cycles. Patients will complete visits on cycle 1 days 1, 4, 8, 15; cycle 2 days 1, 15; day 1 of cycles 3 through 6; and day 1 of every 2 cycles thereafter until discontinued from the program.

An end of treatment visit will be performed within 7 days after last dose of medicinal product (gilteritinib [ASP2215]), or prior to initiation of another anticancer therapy, whichever occurs earlier, followed by a 30-day follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient is considered an adult according to local regulation at the time of signing informed consent.
* Patient has a diagnosis of primary AML or AML secondary to myelodysplastic syndrome or therapy-related AML according to World Health Organization (WHO) classification as determined by pathology review at the treating institution.
* Patient has presence of the FLT3 mutation (internal tandem duplication and/or tyrosine kinase domain [D835/I836] mutation) in bone marrow or peripheral blood.
* Patient has refractory or relapsed AML (with or without Hematopoietic stem cell transplant (HSCT)) or has AML in CRc (CR, CRi, CRp) with Minimal residual disease (MRD) by flow cytometry or genetic testing for the FLT3 mutation after induction/consolidation regimen or HSCT.
* There is no comparable or satisfactory alternative therapy to treat the patient's AML.
* Patient has not received any chemotherapy or investigational agent within at least 5 half-lives after stopping that drug and before starting gilteritinib (ASP2215).
* Patient must meet the following criteria as indicated on clinical laboratory tests:

  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 institutional upper limit of normal
  * Serum total bilirubin ≤ 2.5 mg/dL, except for patients with Gilbert's syndrome
  * Serum potassium and serum magnesium ≥ institutional lower limit of normal.
* Patient is able to tolerate oral administration of gilteritinib (ASP2215).
* Patient who has developed overall grades II-IV acute graft-versus-host disease (GVHD) must satisfy the following criteria:

  * No requirement of > 0.5 mg/kg of prednisone (or equivalent) daily dose within 1 week of the initiation of gilteritinib (ASP2215) treatment.
  * No escalation of immunosuppression in terms of increase of corticosteroids or addition of new agent/modality in prior 2 weeks (note that increasing calcineurin inhibitors or sirolimus to achieve therapeutic trough levels is allowed).
* Female patient must either:

  * Be of nonchildbearing potential: Postmenopausal (defined as at least 1 year without any menses for which there is no other obvious pathological or physiological cause) prior to screening, or Documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 1 month prior to screening
  * Or, if of childbearing potential, agree not to try to become pregnant during the program and for at least 180 days after the final medicinal product administration, and have a negative serum or urine pregnancy test at screening and, if heterosexually active, agree to use consistently 2 forms of effective contraception per locally accepted standards (1 of which must be a barrier method) starting at screening and throughout the program period and for at least 180 days after the final medicinal product administration.
* Female patient must agree not to breastfeed or donate ova starting at screening and throughout the program period, and for at least 180 days after the final medicinal product administration.
* Male patient (even if surgically sterilized) and their partners who are women of childbearing potential must agree to practice 2 forms of effective contraception per locally accepted standards (1 of which must be a barrier method), starting at screening and throughout the program period and for 120 days after the final medicinal product administration.
* Male patient must not donate sperm starting at patient evaluation and throughout the program period and for 120 days after the final medicinal product administration.
* Patient agrees not to participate in an interventional study for AML while on treatment.
* Patient who has a diagnosis of human immunodeficiency virus may be registered in the program as long as their disease is under control on antiretroviral therapy. Precautions should be taken to modify their highly active antiretroviral therapy regimen to minimize drug interactions.

Exclusion Criteria:

* Patient is able to participate in an ongoing clinical study of gilteritinib (ASP2215); or has previously participated in a randomized clinical study of gilteritinib (ASP2215) with a primary endpoint of survival that is not closed for efficacy.
* Patient with Fridericia-corrected QT interval (QTcF) > 450 ms at the screening visit based on local reading.
* Patient with a known history of Long QT Syndrome at the screening visit.
* Patient was diagnosed with acute promyelocytic leukemia (APL).
* Patient has BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Patient has clinically significant coagulation abnormality unless secondary to AML.
* Patient has active hepatitis B or C or an active hepatic disorder.
* Patient has uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia, or New York Heart Association Class IV heart failure.
* Patient requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP) 3A.
* Patient has any condition which makes the patient unsuitable for participation in the program.
* Patient has hypersensitivity to any of the medicinal product components.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (6):
- Site AU61001, Canberra, Australia
- Italy (2):
  - Site IT39001, Milan
  - Site IT39003, Milan
- United Kingdom (3):
  - Site UK44001, Birmingham
  - Site UK44003, Bristol
  - Site UK44002, London

REFERENCES:
- [Derived] Dogu MH, Tekgunduz AIE, Deveci B, Korkmaz G, Comert M, Sevindik OG, Yokus O, Serin I. Gilteritinib (XOSPATA(R)) in Turkey: Early Access Program Results. Mediterr J Hematol Infect Dis. 2023 May 1;15(1):e2023031. doi: 10.4084/MJHID.2023.031. eCollection 2023. PMID 37180209